CLINICAL TRIAL: NCT02175160
Title: Predictability of the Ability to Perform an Emergency Stop in Knee Osteoarthritis and Patients With Total Knee Arthroplasty
Brief Title: Predictability of the Ability to Perform an Emergency Stop
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 619/2013BO2
Record Dates: First submitted 2014-06-11; First posted 2014-06-26 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2014-06

CONDITIONS: Osteoarthritis; Total Knee Arthroplasty
Keywords: Driver reaction time
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Braking and functionality with right knee osteoarthritis (Experimental): Cohort testing of driving performance in a drive simulator and correlation with clinical functionality in patients with right knee osteoarthritis
  Interventions: Other: Braking and functionality
- Braking and functionality with right knee arthroplasty (Experimental): Cohort testing of driving performance in a drive simulator and correlation with clinical functionality in patients with right total knee arthroplasty
  Interventions: Other: Braking and functionality

INTERVENTIONS:
Other: Braking and functionality

SUMMARY:
Several studies exist on patient performance in drive simulators especially around and after surgery. Recommendations concerning the ability to drive preoperatively are based on these studies, which generated their data using drive simulators. However, in all the datasets driving performance remains highly individual. Since a drive simulator is not readily available in normal general practitioner surgeries it would be helpful to have convenient clinical tests to evaluate a patients individual ability to perform an emergency stop. This study aims at evaluating different possibilities how such performance might be predicted. Patients with knee osteoarthritis and patients who have received total knee arthroplasty are tested clinically and their results are compared with the gold standard experiment - a drive simulator.

ELIGIBILITY:
Inclusion Criteria:

* 18-85 y
* valid driving license
* male and female
* right or left knee Osteoarthritis, Total knee arthroplasty right or left knee
* capability to walk with or without a walking stick

Exclusion Criteria:

* myocardial infarction/Apoplexia < 6 months
* Total knee arthroplasty <5 weeks
* New York Heart Association 3/4
* lacking drivers' license
* peripheric sensomotor deficit <3/5 British Medical Research Council
* new fracture of the lower extremity or spine
* systemic or metastasised Cancer
* drug intake with centrally acting substances known to affect reaction time (Opioids, e.g. Tramadol, oxycodone, morphine, Tilidin)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-07; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Correlation of knee functionality and braking performance | Osteoarthritis group: at consultation, Total knee arthroplasty group: more than 5 weeks postoperatively, at consultation
  Evaluation of degree of correlation of braking performance (total brake response time) and clinical testing of knee functionality in patients with right knee osteoarthritis or total knee arthroplasty.
  One time point of evaluation for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Ulf K Hofmann, MD, Principal Investigator — University Hospital Tuebingen
Locations (1):
- University Hospital Tuebingen, Department of Orthopaedics, Tübingen, Germany

REFERENCES:
- [Result] Hau R, Csongvay S, Bartlett J. Driving reaction time after right knee arthroscopy. Knee Surg Sports Traumatol Arthrosc. 2000;8(2):89-92. doi: 10.1007/s001670050192. PMID 10795670